CLINICAL TRIAL: NCT04000022
Title: Comparative Efficacy of Repetitive Transcranial Magnetic Stimulation in Pharmaco-naïve and Treatment Resistant Patients With Major Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation in Pharmaco-naïve Patients With Major Depression
Acronym: NAIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Maximilian Kiebs, M.S. (Unknown); Clemens Mielacher, M.S. (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Head Medical Psychology Division, Vice Head Psychiatry Department, Principal Investigator, Full Professor, University Hospital, Bonn
Other Study IDs: NAIV
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; rTMS; TBS; Theta Burst Stimulation; Neuronavigation; Non-Treatment Resistant; Pharmaco-Naïve
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Non-Treatment Resistant Patients
  Interventions: Device: intermittent theta burst stimulation (iTBS)
- Treatment-Resistant Patients: The group of patients from NCT03944213
  Interventions: Device: intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) — 20 sessions of iTBS

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has become a safe and efficacious treatment for patients with treatment-resistant depression. In several studies investigating the antidepressant efficacy of rTMS, it has been shown that in low treatment-resistant patients rTMS is more efficacious than in patients where several treatment attempts have failed. Albeit this finding, most studies to date primarily recruited patients with relatively high degrees of treatment-resistance and there is a lack of trials investigating rTMS as a first-line treatment. Therefore, this trials aims to compare the antidepressant efficacy of 4 weeks open-label theta-burst TMS in non-treatment-resistant patients with a comparable group of treatment-resistant MDD patients.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) has become a safe and efficacious treatment for patients with treatment-resistant depression (Mutz et al., 2019). Consequently, several countries including Australia, Brazil, Canada, Israel and the United States have approved rTMS as second-line treatment for major depressive disorder (MDD), while others have included rTMS in their guidelines for good clinical practice (e.g. Finland, Germany and Serbia). Historically, rTMS was conceptualized as a "soft" alternative to electroconvulsive therapy. Therefore, most studies to date primarily recruited patients with relatively high degrees of treatment-resistance (> two failed treatment attempts) and there is a lack of trials investigating rTMS as a first or second line treatment. This finding is contrasted by the fact that on the most stable predictors of response to rTMS is low-treatment resistance.

Therefore, this trial aims to compare the antidepressant efficacy of 20 pharmaco-naïve patients with 20 treatment-resistant patients diagnosed with major depressive disorder. In this open label trial, patients will receive four weeks high-frequency left-sided theta burst TMS (lDLFPC). The target will be located by neuronavigation to the target ascertained by Fox et al.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to provide consent.
* Diagnosis of Major Depressive Disorder according to DSM-V criteria.
* The duration of the current episode is at least four weeks and no more than five years.
* During the current episode, pharmacological intervention was prescribed (and taken) by the patient

Exclusion Criteria:

* The participant does not fulfill requirements for iTBS treatment according to safety guidelines.
* Cardiac or neurological surgery, active implants, metal parts within the body, claustrophobia.
* Pregnancy or breast-feeding.
* Psychiatric illness, e.g. substance abuse, psychosis, bipolar disorder, anorexia, obsessive compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder, personality disorder.
* Antipsychotic medication not approved for the treatment of depression.
* Acute suicidality.
* Conditions related to increased intracranial pressure.
* Brain injury or stroke.
* History of epilepsy in patient or in first-degree relative.
* Cerebral aneurysm.
* Neurological illness (e.g. dementia (score of less than 25 in Mini Mental State Exam), Parkinson's disease, chorea huntington, multiple sclerosis).
* Course of electroconvulsive therapy (ECT) within the last three months

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients at the psychiatric hospital of the University Hospital Bonn. The patients diagnosis of major depressive disorder will be verified via the structured clinical interview for DSM-5. iTBS protocols in line with international standards administered by a trained professional.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression severity as measured by the Hamilton Depression Rating Scale (HDRS-17) over 7 timepoints | Six weekly measurements starting 1 week before first iTBS treatment session, one follow-up measurement four weeks after last measurement
  Remission defined as HDRS-17 score (range: 0 to 52) of less than or equal to 8 after the iTBS course. Response defined as a reduction of at least 50% from baseline in HDRS-17 score after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fregni F, Marcolin MA, Myczkowski M, Amiaz R, Hasey G, Rumi DO, Rosa M, Rigonatti SP, Camprodon J, Walpoth M, Heaslip J, Grunhaus L, Hausmann A, Pascual-Leone A. Predictors of antidepressant response in clinical trials of transcranial magnetic stimulation. Int J Neuropsychopharmacol. 2006 Dec;9(6):641-54. doi: 10.1017/S1461145705006280. Epub 2005 Nov 23. PMID 16939662
- [Background] Brakemeier EL, Luborzewski A, Danker-Hopfe H, Kathmann N, Bajbouj M. Positive predictors for antidepressive response to prefrontal repetitive transcranial magnetic stimulation (rTMS). J Psychiatr Res. 2007 Aug;41(5):395-403. doi: 10.1016/j.jpsychires.2006.01.013. Epub 2006 Mar 22. PMID 16554071
- [Background] Lisanby SH, Husain MM, Rosenquist PB, Maixner D, Gutierrez R, Krystal A, Gilmer W, Marangell LB, Aaronson S, Daskalakis ZJ, Canterbury R, Richelson E, Sackeim HA, George MS. Daily left prefrontal repetitive transcranial magnetic stimulation in the acute treatment of major depression: clinical predictors of outcome in a multisite, randomized controlled clinical trial. Neuropsychopharmacology. 2009 Jan;34(2):522-34. doi: 10.1038/npp.2008.118. Epub 2008 Aug 13. PMID 18704101
- [Background] Mutz J, Vipulananthan V, Carter B, Hurlemann R, Fu CHY, Young AH. Comparative efficacy and acceptability of non-surgical brain stimulation for the acute treatment of major depressive episodes in adults: systematic review and network meta-analysis. BMJ. 2019 Mar 27;364:l1079. doi: 10.1136/bmj.l1079. PMID 30917990
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Kiebs M, Hurlemann R, Mutz J. Repetitive transcranial magnetic stimulation in non-treatment-resistant depression. Br J Psychiatry. 2019 Aug;215(2):445-446. doi: 10.1192/bjp.2019.75. Epub 2019 Apr 24. PMID 31014413